CLINICAL TRIAL: NCT06636526
Title: The i4i PRODICT® Study: Evaluation of the i4i PRODICT® Test in Different Ethnic Groups.
Brief Title: The i4i PRODICT® Study: Evaluation of the i4i PRODICT® Test in Different Ethnic Groups (The i4i PRODICT® Study).
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CCR6045
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate cancer screening; Polygenic risk score; PSA; Genetic Predisposition
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Risk Score; Genetic Predisposition to Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood & urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1: People with a prostate aged 40-55 years of either (i) Black African and Black African-Caribbean, (ii) South Asian or East Asian or (iii) White European ancestry to undergo genetic testing using the i4i PRODICT® test to identify those at higher genetic risk for prostate cancer targeted screening.
  Interventions: Genetic: The i4i PRODICT® test.
- Part 2: Those classified as high-risk due to either falling within the high polygenic risk score category, and/or having a rare variant in a gene in the i4i PRODICT® test will be offered a hospital clinic appointment at the Royal Marsden Hospital to discuss prostate cancer screening.
  Interventions: Genetic: The i4i PRODICT® test.; Other: Prostate cancer screening; Procedure: MRI Scan; Procedure: Prostate Biopsy

INTERVENTIONS:
Genetic: The i4i PRODICT® test. — The i4i PRODICT® test combining both common and rare genetic variants into one saliva-based DNA test to estimate a person's future risk of prostate cancer. This test will be offered to all participants in Part 1 of the study. Participants will be classified into high-risk or population risk based on the results of the i4i PRODICT® test. Those classified as high-risk due to either falling within the high polygenic risk score category, and/or having a rare variant in a gene in the test will be offered targeted prostate cancer screening.
Other: Prostate cancer screening — Prostate cancer screening in the form of PSA testing will be offered to all participants identified as high risk from the i4i PRODICT® test for three years in order to track development of cancer in the future.
  Groups: Part 2
Procedure: MRI Scan — MRI scan will be offered to participants identified in the high-risk category of the i4i PRODICT® test depending on their PSA test results. Where PSA is above age-specific threshold (>2.5ug/L for people with prostates (PwPs) aged 40-50 years and >3.5ug/L for PwPs aged 50-55 years), those with raised PSA levels will be referred for multiparametric MRI at The Royal Marsden Hospital.
  Groups: Part 2
Procedure: Prostate Biopsy — Transperineal prostate biopsy under local anaesthetic will be offered to to participants identified in the high-risk category of the i4i PRODICT® test depending on their MRI results. Where a lesion is visible on MRI (defined as a PIRAD score ≥3) onward referral will be made for a transperineal targeted prostate biopsy (or current gold standard NHS practice).
  Groups: Part 2

SUMMARY:
The i4i PRODICT® study has been developed to investigate the uptake and acceptability of the i4i PRODICT® test which combines both common and rare genetic changes (genetic variants) into one saliva-based DNA test to estimate a person's future risk of prostate cancer (PrCa) in people of varying ethnicities.

DETAILED DESCRIPTION:
The i4i PRODICT® study aims to recruit 1000 people with a prostate (PwP*) aged 40-55 years old, divided into three ethnic backgrounds: (i) Black African and Black African-Caribbean, (ii) South Asian or East Asian or (iii) White European ancestry. These ethnic backgrounds are defined as having all 4 grandparents of the same ancestry. *People with a prostate is defined as people born male. We believe this will provide us with data that are reproducible and implementable within the UK population as well as enrich recruitment from underserved non-White European communities in order to evaluate this approach within a future potential national screening programme.

Recruitment is taking place via collaborating General Practice (GP) surgeries. For recruitment via GP practices, potential participants will be contacted via a letter from their GP, including a Participant Information Sheet (PIS) and if interested in the study, they will be asked to complete a reply slip found at the back of the PIS and return it to the study team for further information. Potential participants will also be identified through advertisements in the press, use of social media (in collaboration with press offices of the ICR/RMH, the funders of the study), outreach work in communities, presentations, posters/leaflets and animation videos about the study that could be displayed in GP surgeries, hospitals, public spaces and other community organisations. Potential participants identified via these routes will be considered as direct expressions of interest. For recruitment via direct expression of interest, potential participants can contact the study team directly to express interest in taking part in this study and receive further information. All potential participants will be sent a consent form and an eligibility questionnaire for completion.

Consented eligible participants will then be sent a DNA collection saliva kit. DNA will be extracted from saliva and analysed using the i4i PRODICT® test. Those participants identified at higher genetic risk (corresponding to the top 20% of the White European cohort, top 50% of the Black African/ African-Caribbean cohort and top 10% of the Asian cohort or those identified as having a rare variant) will be invited for prostate cancer (PrCa) screening annually for 3 years at the Royal Marsden Hospital. PrCa screening will mirror the primary care pathway: those in the high-risk group will be offered a PSA test and managed according to age-appropriate PSA thresholds. Where indicated, onward referral for prostate MRI, and prostate biopsy will follow as per the National Institute for Health and Care Excellence (NICE) guidelines. For participants receiving a diagnosis of PrCa, they will be offered treatment at The Royal Marsden Hospital, or onward referral to their local cancer centre if preferred by the patient.

ELIGIBILITY:
Inclusion Criteria:

* People with a prostate* (PwP). *People with a prostate is defined as people born male.
* Aged 40 to 55 years.
* People of either (i) Black African/Black African-Caribbean; (ii) White European; or (iii) South Asian or East Asian ancestry. These are defined as individuals with 4 grandparents of the same ancestry.
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Previous diagnosis of prostate cancer.
* People of mixed ancestry
* Previous diagnosis of cancer with a life-expectancy of less than five years.
* Negative prostate biopsy within one year before recruitment.
* Any significant psychological conditions that may be worsened or exacerbated by participation in the study.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The i4i PRODICT® study will be open to people with a prostate* (PwP). *People with a prostate is defined as people born male.
Study Population: People with a prostate* (*defined as people born male), aged 40 - 55 years old of either (i) Black African and Black African-Caribbean, (ii) South Asian or East Asian or (iii) White European ancestry willing to undergo the i4i PRODICT® test to identify those at higher genetic risk for prostate cancer targeted screening.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2033-01-06 (Estimated)

PRIMARY OUTCOMES:
The number of participants stratified by each ethnic background recruited and risk stratified using the i4i PRODICT® test. | 2 years
  Total recruitment target is 1000 participants, split between three ethnic groups: Black African/Caribbean, South Asian and White.

SECONDARY OUTCOMES:
Calculation of the incidence of prostate cancers in the study population. | 3 years
  Calculation of incidence, reported as number of cancers, and percentage incidence of the study population.
Record of clinical features of cancers diagnosed using the NCCN prostate cancer classification system | 8 years
  To look at clinical features and features of aggressiveness of the cancers diagnosed in the study population for comparison with general population data reporting clinical features of cancers diagnosed through routine diagnostic pathways.
Calculation of the proportion of individuals taking up the study stratified by ethnic group. | 1 year
  To look at whether there is equal recruitment across all target ethnic groups
Calculation of the attrition rate stratified by ethnic group. | 3 years
  Understand whether there are differences in attrition in different groups
Number of participants who comply with all components of the study protocol stratified by ethnic group. | 3 years
  To understand whether there are differences in protocol compliance in different groups
Identification of barriers to protocol implementation | 3 years
  Using qualitative research methods barriers to the implementation of the protocol will be identified to inform implementation into routine healthcare

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP; FRCR, Principal Investigator — The Institute of Cancer Research and The Royal Marsden NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - The Institute of Cancer Research and The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden Hospital, London
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the study Steerning Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Within 18 months of the study opening the study protocol will be published
Access Criteria: Study protocol will be published in a peer review journal. For access to other study documents an application can be made to the Steering Committee